CLINICAL TRIAL: NCT00640770
Title: A Prospective, Randomized, Multicenter Comparison of Balloon Angioplasty and the Cypher Selecttm + Coronary and Infrapopliteal Stent in the Treatment of Subjects With Ischemic Infrapopliteal Arterial Disease
Brief Title: Comparing Angioplasty and DES in the Treatment of Subjects With Ischemic Infrapopliteal Arterial Disease
Acronym: ACHILLES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Hans-Peter Stoll - MD, PhD - Worldwide VP Clinical Research & Operations, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EE06-02
Record Dates: First submitted 2008-03-14; First posted 2008-03-21 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Peripheral Arterial Diseases
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon; Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- balloon angioplasty (Active Comparator): balloon angioplasty
  Interventions: Device: balloon angioplasty
- Drug eluting stent (Experimental): CYPHER SELECT+ Coronary or Infrapopliteal Stent
  Interventions: Device: drug eluting stent

INTERVENTIONS:
Device: balloon angioplasty — balloon angioplasty
  Arms: balloon angioplasty
Device: drug eluting stent — Cypher Select+ Coronary or Infrapopliteal Stent
  Arms: Drug eluting stent

SUMMARY:
The primary objective of this study is to compare the performance of the CYPHER SELECTTM + Sirolimus-eluting Balloon-expandable Coronary and Infrapopliteal Stent over balloon angioplasty in de novo and restenotic native below the knee tibioperoneal, anterior and/or posterior tibial and/or peroneal arterial lesions in a prospective, multicenter, randomized clinical study.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized study to be conducted in 18 centers in Europe. A total of 200 subjects will be entered into the study and will be randomized on a 1:1 basis to either balloon angioplasty or the CYPHER SELECTTM + Coronary and Infrapopliteal Stent for infrapopliteal use in subjects with symptomatic peripheral artery disease (Rutherford 3, 4, or 5).

All subjects will undergo a repeat angiography at 12 months to assess the primary endpoint of In-Segment Binary Restenosis. Follow-up visits are scheduled at 6 weeks, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >= 18 and <= 85 years old;
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation;
* Clinical diagnosis of symptomatic critical limb ischemia as defined by Rutherford 3, 4, or 5;
* Single treatment of de novo or restenotic (after PTA only) lesion(s) in the tibioperoneal trunk, anterior and/or posterior tibial and/or peroneal artery;
* A maximum of 2 vessels in 1 limb may be treated in the study, each vessel for only 1 target lesion, resulting in at single risk target lesion(s); In case 1 target lesion is located in the Tibioperoneal trunk, the 2nd target lesion (if applicable) can only be located in the anterior tibial artery; Additional non-target lesion(s) in remaining non-target vessel(s) can be treated at the physician's discretion by means of balloon dilation (± bail-out stenting);
* The sum of the total length of both target lesions can be maximum 120 mm;
* In total a maximum of 4 stents may be implanted to fully cover the maximum of 2 target lesions per subject;
* Target vessel is >= 2.5 and <= 3.5 mm in diameter (visual estimate);
* Target lesion stenosis is >70% diameter stenosis (visual estimate);
* Guidewire must be across the first (if applicable) target lesion and located intraluminally within the distal vessel before study randomization;
* Willing to comply with the specified follow-up evaluation;
* Written informed consent prior to any study procedures.

Exclusion Criteria:

* Significant (>50%) stenoses distal to the target lesion that might require revascularization, or impede runoff;
* Angiographic evidence of thrombus within target vessel;
* Thrombolysis within 72 hours prior to the index procedure;
* Lesions not suitable for stenting;
* Lesions (defined as stenosis > 75%) in the common or external iliac, common or superficial femoral and popliteal artery. However, intervention in TASC A and B lesions (max. 15cm) to restore adequate blood flow, in the same index procedure is allowed. This intervention must be prior to the treatment of the study lesion(s) and successful;
* Lesions located at the bifurcation requiring treatment of both branches (1 in main branch and 1 in side branch);
* Required stent placement across or within 1 cm of the knee joint; in an artery subject to external compression, or in an artery directly subject to movement of the ankle or knee joint;
* Prior stent(s) within the target vessel(s);
* Aneurysm in the SFA or popliteal artery;
* Requiring popliteal arterial access;
* Concomitant hepatic insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy;
* Recent MI or stroke < 30 days prior to the index procedure;
* Coronary intervention < 30 days prior to the index procedure;
* Life expectancy less than 12 months;
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb;
* Impaired renal function (creatinine > 2.5 mg/dl);
* Known or suspected allergies or contraindications to aspirin, clopidogrel bisulfate (PlavixÒ) and ticlopidine (Ticlidâ), heparin, stainless steel or contrast agent;
* The subject is currently taking Coumarin / Warfarin which, in the opinion of the investigator, interferes with the subject's participation in the study;
* Any significant medical condition which, in the investigator's opinion, may interfere with the subject's optimal participation in the study;
* The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
In-Segment Binary Restenosis | 12-months

SECONDARY OUTCOMES:
Mean percent diameter stenosis (%DS) and minimal lumen diameter (MLD) measured by quantitative angiography post-procedure. | 12 months
In-segment late loss measured by quantitative angiography. | 12 months
In-stent late loss measured by quantitative angiography. | 12 months
Patency defined as detectable flow measured by Duplex Ultrasound. | 6 weeks, 6 and 12 months
Target Lesion Revascularization (TLR), and Target Vessel Revascularization (TVR). | 6 weeks, 6 and 12 months;
Assessment for stent fractures by X-Ray. | 12 months
Device Success defined as achievement of a final residual diameter stenosis of <30% (by QA), using the assigned device only. | post procedure
Lesion Success defined as achievement of <50% (by QA) residual stenosis using any percutaneous method. | post procedure
Procedural Success defined as achievement of final diameter stenosis of <50% (by QA) using any percutaneous method, without the occurrence of an SAE up to catheter sheath removal or subject leaving the cath lab, whichever is earlier. | post procedure
Procedural Complications defined as any adverse event from the time of arterial punction up to the moment of catheter sheath removal or subject leaving the cath lab, whichever is earlier. | post procedure
Serious Adverse Events | At procedure up to discharge, 6 weeks, 6 and 12 months
Rutherford classification | At screening, 6 weeks, 6 and 12 months
Ankle Brachial Index measured | At screening, 6 weeks, 6 and 12 months
Amputation | 6 weeks, 6 and 12 months
Quality of Life assessment. | 6 weeks, 6 and 12 months
Wound status of index limb (if applicable) due to CLI measured by digital photography, depth/length/width measurements, infection and wound closure status. | screening, 6 weeks, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, PhD, Principal Investigator — Universität Leipzig - Herzzentrum
Locations (1):
- Universität Leipzig - Herzzentrum, Leipzig, Germany

REFERENCES:
- [Derived] Katsanos K, Spiliopoulos S, Diamantopoulos A, Siablis D, Karnabatidis D, Scheinert D. Wound Healing Outcomes and Health-Related Quality-of-Life Changes in the ACHILLES Trial: 1-Year Results From a Prospective Randomized Controlled Trial of Infrapopliteal Balloon Angioplasty Versus Sirolimus-Eluting Stenting in Patients With Ischemic Peripheral Arterial Disease. JACC Cardiovasc Interv. 2016 Feb 8;9(3):259-267. doi: 10.1016/j.jcin.2015.10.038. Epub 2016 Jan 6. PMID 26777329